CLINICAL TRIAL: NCT03120897
Title: Rainbow Acoustic Monitoring (RAM) Clinical Engineering Data Collection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision to terminate study.
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DROV0008
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test group (Experimental): The subjects will be enrolled into the test group and will receive RAM sensor.
  Interventions: Device: RAM sensor

INTERVENTIONS:
Device: RAM sensor — Rainbow Acoustic Monitoring sensor for measurement of respiratory rate

SUMMARY:
To capture high resolution waveform data and numerical data from investigational and FDA-released RAM sensors in the neonatal, infant, pediatric, and adult patient population

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects that are between 0 to 70 years old.
* Neonate, Infant, Pediatric, Adult, and Pregnant subjects with fully developed skin.

Exclusion Criteria:

* Patients with skin abnormalities at the planned application sites that would interfere with sensor, cannula or electrode applications.
* Patients with pre-existing conditions and/or co-morbidities that would prohibit them from participating in the study due to unacceptable risks to their health and well-being, as determined by the Principal Investigator (PI).
* Patients who the PI deems ineligible at the PI's discretion

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-06; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects in which respiratory rate is collected | Duration of surgery
  Capture high resolution waveform data and numerical data from respiratory rate using RAM sensor

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Medical Center, Stanford, California, United States